CLINICAL TRIAL: NCT06452693
Title: A Phase Ib/IIa Clinical Trial to Evaluate the Safety, Tolerability, Pharmacokinetic, and Antiviral Efficacy of TQA3038 Injection in Patients With Chronic Hepatitis B
Brief Title: A Clinical Study to Evaluate the Efficacy of TQA3038 Injection in Patients With Chronic Hepatitis B
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TQA3038-Ib/IIa-01
Record Dates: First submitted 2024-06-06; First posted 2024-06-11 (Actual); Last update posted 2024-06-11 (Actual); Status verified 2024-03

CONDITIONS: Hepatitis B, Chronic
MeSH Terms: conditions — Hepatitis B, Chronic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TQA3038 injection/placebo (Experimental): 100/0mg~400/0mg, subcutaneous injection, 2 weeks~8 weeks as a cycle, a total of 2 doses.
  Nucleotide drugs: Oral, once a day, orally administered with food, for 16 weeks.
  Interventions: Drug: TQA3038 injection/placebo
- Nucleotide drugs Control group (Active Comparator): Nucleotide drugs: Oral, once a day, orally administered with food, for 48weeks.
  Interventions: Drug: Nucleotide drugs Control group

INTERVENTIONS:
Drug: TQA3038 injection/placebo — TQA3038 is a Anti-Hepatitis B virus (HBV) drugs.
  Arms: TQA3038 injection/placebo
Drug: Nucleotide drugs Control group — Nucleotide drugs are nucleoside reverse transcriptase inhibitors.
  Arms: Nucleotide drugs Control group

SUMMARY:
This study is divided into two parts. Phase Ib is a randomized, double-blind, placebo-controlled trial, designed to evaluate the safety, tolerability, pharmacokinetic characteristics, preliminary efficacy, and immunogenicity of TQA3038 injection in patients with chronic hepatitis B. It is expected to include 72 subjects. Phase IIa adopted an open-label, randomized, parallel-controlled design, with a total of 90 subjects included, mainly evaluating the changes in serum HBsAg compared to baseline at the end of the 48th week.

ELIGIBILITY:
Inclusion Criteria:

* Subjects voluntarily participate in this study and sign informed consent;
* Male and female ≥18 years old and ≤65 years old;
* Male subjects with a weight of ≥ 50 kilograms and female subjects with a weight of ≥ 45 kilograms, BMI 18~28 kg/m2;
* Patients diagnosed with chronic hepatitis B (CHB) who have been serum HBsAg positive for more than 6 months and HBeAg positive ; During the screening period, 100 IU/ml ≤ HBsAg quantification ≤ 5000 IU/ml;
* The subjects are able to communicate well with the researchers, voluntarily and can understand and follow the experimental protocol process to complete the study;
* The subjects (including partners) are willing to voluntarily adopt effective contraceptive measures during the clinical trial period and long-term follow-up period, and specific contraceptive measures are shown in the appendix;
* The treated patients need to meet the condition:The subject must have received oral nucleoside (acid) drug treatment and a stable treatment regimen;
* Newly treated patients must meet the condition:During screening, the subjects had never received antiviral treatment for chronic hepatitis B B (oral nucleoside (acid) drugs and interferon), or had irregular antiviral treatment in the past, but had not received any antiviral treatment for chronic hepatitis B 3 months before enrollment.

Exclusion Criteria:

* Pregnant and lactating women;
* Chronic diseases other than chronic HBV infection with significant clinical significance that have a history of mental illness or are deemed unsuitable by researchers for participation in this study;
* Acute diseases with significant clinical significance occurring within 7 days prior to receiving the investigational drug;
* Individuals with a history of active pathological bleeding or a tendency towards bleeding;
* Prescription medication has been used within 14 days prior to receiving the study drug;
* Receive any preventive or attenuated vaccines within 14 days prior to receiving the study drug;
* Blood donors or those who have lost a significant amount of blood within the first 3 months of screening, or those who have donated blood during the planned study period;
* Subjects with a history of excessive alcohol consumption;
* A history of alcohol or drug abuse within the 12 months prior to screening, or a positive drug screening result during screening;
* Complicated with other infected disease;
* Patients with significant liver fibrosis or cirrhosis before or during screening;
* History of chronic liver diseases other than chronic HBV infection;
* Patients have a history of hepatocellular carcinoma (HCC) before or at the time of screening, or may be at risk for HCC;
* Used immunosuppressive or immunomodulatory drugs and cytotoxic drugs within 6 months prior to the study medication;
* During screening, subjects showed significant laboratory results abnormalities；
* Screening for tumors with a history of malignancy within the first 5 years, excluding tumors that can be completely cured through surgical resection;
* Uncontrollable chronic diseases;
* History of intolerance to subcutaneous injection;
* Participated in clinical studies of any drug or medical device within 3 months prior to drug administration or within 5 times the half-life of the investigational drug, or used the investigational drug;
* Those considered unsuitable for enrollment by the investigators.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 162 (Estimated)
Dates: Start 2024-06 (Estimated); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Adverse events (AEs) | Baseline up to 16 weeks
  The incidence of adverse events (AEs) during treatment.
Serious adverse events (SAEs) | Baseline up to 16 weeks
  The incidence of serious adverse events (SAEs) during treatment.
Hepatitis B virus surface antigen (HbsAg) | Baseline up to 48 weeks
  Changes of serum HbsAg compared with baseline at the 48th week of treatment in each group.

SECONDARY OUTCOMES:
Time to Reach Maximum Plasma Concentration (Tmax) | Predose on the 1st dose administration and 30 minutes, 1, 2, 4, 8, 24hours postdose and Predose on the 2nd dose administration and 30 minutes, 1, 2, 4, 8, 24hours postdose
  Time to reach Cmax of TQA3038 and its metabolite in plasma.
Maximum Plasma Concentration (Cmax) | Predose on the 1st dose administration and 30 minutes, 1, 2, 4, 8, 24hours postdose and Predose on the 2nd dose administration and 30 minutes, 1, 2, 4, 8, 24hours postdose
  Maximum concentration of TQA3038 and its metabolite in plasma.
Area Under the Plasma Concentration Versus Time Curve (AUC) | Predose on the 1st dose administration and 30 minutes, 1, 2, 4, 8, 24hours postdose and Predose on the 2nd dose administration and 30 minutes, 1, 2, 4, 8, 24hours postdose
  Area under the curve of TQA3038 and its metabolite from time 0 to last measurable time.
Volume of distribution (Vd/F) | Predose on the 1st dose administration and 30 minutes, 1, 2, 4, 8, 24hours postdose and Predose on the 2nd dose administration and 30 minutes, 1, 2, 4, 8, 24hours postdose
  Volume of distribution (Vd/F) of TQA3038 in Plasma.
Apparent Plasma Clearance (CL/F) | Predose on the 1st dose administration and 30 minutes, 1, 2, 4, 8, 24hours postdose and Predose on the 2nd dose administration and 30 minutes, 1, 2, 4, 8, 24hours postdose
  Apparent Plasma Clearance (CL/F) of TQA3038 in Plasma.
Apparent Terminal Elimination Half-life (t1/2) | Predose on the 1st dose administration and 30 minutes, 1, 2, 4, 8, 24hours postdose and Predose on the 2nd dose administration and 30 minutes, 1, 2, 4, 8, 24hours postdose
  Apparent Elimination Half-life (T1/2) of TQA3038 in Plasma
The incidence and titer of anti drug antibodies (ADA) | Day1 before administration, Week 8, Week 16, and during withdrawal
  The incidence and titer of anti drug antibodies (ADA) in serum.
Incidence of Neutralization antibody (Nab) | Day1 before administration, Week 8, Week 16, and during withdrawal
  Incidence of Neutralization antibody (Nab) in serum.
Hepatitis B surface antigen (HBsAg) | Baseline up to 48 weeks
  Changes in Hepatitis B surface antigen (HbsAg) levels from baseline during the study period.
Hepatitis B E antigen (HBeAg) | Baseline up to 48 weeks
  Changes in HbeAg levels from baseline during the study period.

CONTACTS AND LOCATIONS:
Locations (22):
- China (22):
  - The First Affiliated Hospital of Bengbu Medical College, Bengbu, Anhui
  - Mengchao Hepatobiliary Hospital of Fujian Medical University, Fuzhou, Fujian
  - Gansu province people hospital, Lanzhou, Gansu
  - The Third Affiliated Hospital of Sun Yat sen University, Guangzhou, Guangdong
  - The First Affiliated Hospital of GUANGXI Medical University, Nanning, Guangxi
  - Guizhou Provincial People's Hospital, Guiyang, Guizhou
  - The Fourth Affiliated Hospital of Harbin Medical University, Harbin, Heilongjiang
  - Shiyan City Taihe Hospital, Shiyan, Hubei
  - Tongji Hospital of Tongji medical college of HUST, Wuhan, Hubei
  - Xiangya Third Hospital of Central of Central Suoth University, Changsha, Hunan
  - The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - The first hospital of Jilin University, Changchun, Jilin
  - Hepatobiliary Hospital of Jilin, Changchun, Jilin
  - The sixth people's hospital at of Shenyang, Shenyang, Liaoning
  - Shengjing Hospital Affiliated to China Medical University, Shenyang, Liaoning
  - Shandong Public Health Clinical Center, Jinan, Shandong
  - West China Hospital of Sichuan University, Chengdu, Sichuan
  - The First Affiliated Hospital of Xinjiang Medical University, Ürümqi, Xinjiang
  - The Southwest Hospital of AMU, Chongqing
  - The Second Affilated Hospital of Chongqing medical university, Chongqing
  - Shanghai Tongren Hospital, Shanghai
  - People's Hospital of Tianjin (City), Tianjin